CLINICAL TRIAL: NCT00272974
Title: Measuring the Impact of Male and Female Condom Promotion Among Commercial Sex Workers in Madagascar
Brief Title: Madagascar Female Condom Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Ministry of Health, Madagascar (Other Government); National Reference Laboratory, Madagascar (Other); University of North Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9713
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2003-08

CONDITIONS: Sexually Transmitted Diseases
Keywords: AE adverse event; DCF data collection forms; IRB Institutional Review Board; SAE serious adverse event
MeSH Terms: conditions — Sexually Transmitted Diseases

INTERVENTIONS:
Behavioral: Clinic-based counseling

SUMMARY:
The study was designed to measure the effects of male and female condom promotion on STI prevalence and reported condom use by sex workers and their partners. It also examined whether the intensity of the education and support given to intended users affected adoption and sustained use of these methods.

The primary objective of the study was:

1. To test the effect of supplementing community-based male and female condom promotion with clinic-based counseling, measured in terms of the level of protection in high-risk sex acts and STI prevalence.

   Secondary objectives of the study included:
2. To monitor short- and medium terms changes in the proportion of protected sex acts among commercial sex workers after the female condom is added to a male condom distribution system.
3. To examine short-term and medium-term changes in STI prevalence when the female condom is added to the male condom distribution system.
4. To measure the incremental cost-effectiveness of adding female condom promotion to existing male condom distribution systems

DETAILED DESCRIPTION:
This three-phased study examined ways to improve services for the prevention of STIs among commercial sex workers. This study was conducted in identical fashion in two sites (Tamatave and Antananarivo) in Madagascar. It tested whether condom promotion through community-based counseling or clinic based counseling leads to an increased level of protection among high-risk sex acts and a subsequent decrease in STI infection rates.

In Phase I, women at each site were randomly assigned to a study arm receiving a community-based male condom promotion intervention, or a study arm receiving community-based male condom promotion supplemented with clinic-based counseling. Randomization was accomplished by the use of sequentially-numbered sealed, opaque envelopes containing the group assignment. The randomization list was stratified by study site. Phase I began with baseline measurement of male condom use and STI prevalence. Participants returned three times, at two month intervals, for follow-up. At each visit, face-to-face interviews were conducted to estimate the proportion of protected sex acts. At the third visit only, participants were tested for gonococcal, chlamydial, and trichomonal infections. This reliance on a combination of biologic and behavioral outcomes helped to reduce any bias brought on by the inherent limitations of either of these measures on its own.

Half the women completing Phase I at each site were then randomized to a Phase II study arm receiving a community-based male and female condom promotion intervention, while the other half entered Phase II receiving the same community-based male and female condom promotion supplemented with clinic-based counseling. This sequential randomization scheme allowed measurement of the short-term (within 6 months) effect of clinic-based counseling on male condom use and STI prevalence, and the short-term effect of clinic-based counseling on male condom + female condom use and STI prevalence. A similar data collection process was used, with measurement of male and female condom use in all three visits, and STI testing in the third visit only.

In Phase III, participants were followed for an additional 6 months, in the same intervention group to which they were assigned at the beginning of Phase II, to assess the medium-term impacts of the female condom, after participants had a chance to become accustomed to the female condom.

ELIGIBILITY:
Inclusion Criteria: Adult female sex workers from the two sites

Exclusion Criteria: None specified

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2001-02; Study Completion 2003-08

PRIMARY OUTCOMES:
Use of protection (male and female condoms)
STIs

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Hatzell, PhD, MPH, Study Chair — FHI 360; Paul Feldblum, PhD, Study Director — FHI 360; Kathleen Van Damme, MD, Principal Investigator — FHI 360
Locations (2):
- Madagascar (2):
  - Isotry Health Center, Antananarivo
  - Dispensaire Kelly, Toamasina

REFERENCES:
- See also: Related Info — http://www.fhi.org